CLINICAL TRIAL: NCT01706601
Title: Patients With Hemorrhoids Referred to a Surgical Specialist Department
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Solveig Elmér, MD, Karolinska Institutet
Other Study IDs: 2010/1108-31/1
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemorrhoids: Patient with hemorrhoids

SUMMARY:
Hemorrhoids is the most common disease in rectum with a prevalence of 30 % of population. This means that many patients are referred to surgical specialist reception with diagnosis hemorrhoidal disease. The aim of this study is to describe population of patients with hemorrhoidal disease that are referred to a specialised colorectal unit and to determine what treatment they are given at a general practitioner as well as in colorectal unit.

ELIGIBILITY:
Inclusion Criteria:

* all patients with diagnosis hemorrhoidal disease that are referred to a surgical specialist department

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whith hemorrhoids
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Correct diagnosis? | patients visiting Ersta Hospital between 2007-2009

SECONDARY OUTCOMES:
treatment of hemorrhoids | patients visiting Ersta Hospital between 2007-2009
  Surgical or conservative treatment, results and number of patients in the groups

OTHER OUTCOMES:
Examination/treatment | Before visiting Ersta hospital
  Examination and treatment given by general practitioner
Operation/complication | postoperatively
  Which operations were performed, complications?, reinterventions?
genus | between 2007-2009
  Did men and women got the same treatment
Treated elsewhere | after compleated treatment at Ersta hospital

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Elmér, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta hospital, Stockholm, Sweden